CLINICAL TRIAL: NCT04899232
Title: Antithrombin III (AT3) in Infectious Disease Caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-COV-2)/ Coronavirus Disease of 2019 (COVID-19)
Brief Title: Antithrombin III in Infectious Disease Caused by COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There are fewer potential patients and an early conclusion of the study would be beneficial in an attempt to finish in a reasonable time and keep the cohorts homogenous.
Sponsor: Enrique Ginzburg (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor-Investigator, Enrique Ginzburg, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20201048
Record Dates: First submitted 2021-05-20; First posted 2021-05-24 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Antithrombin III Deficiency; Covid19
MeSH Terms: conditions — Antithrombin III Deficiency; COVID-19 | interventions — Antithrombin III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- AT3 less than 100% with SOC plus AT3 supplement (Experimental): Participants in this group, with endogenous Antithrombin lll less than 100%, will receive 5 doses of supplemental Antithrombin III on Days 1, 3, 5, 7 and 9, in addition to standard of care (SOC) treatment.
  Interventions: Drug: Antithrombin III
- AT3 less than 100% with SOC only (No Intervention): Participants in this group, with endogenous Antithrombin III less than 100%, will receive SOC treatment only.
- AT3 more than 100% with SOC only (No Intervention): Participants in this group, with endogenous Antithrombin III more than 100%, will receive SOC treatment only.

INTERVENTIONS:
Drug: Antithrombin III — Five total doses of daily 1,821 to 9,100 IUs Antithrombin III, depending on participant's weight, will be administered intravenously every other infusion day (Days 1, 3, 5, 7 and 9).
  Other Names: Thrombate III
  Arms: AT3 less than 100% with SOC plus AT3 supplement

SUMMARY:
The purpose of this research study is to see if participants who have SARS-CoV-2 and low levels of AT3 in the blood will benefit by being given AT3.

ELIGIBILITY:
INCLUSION CRITERIA:

1. >18y of age,
2. Subject or proxy who can provide informed consent
3. Positive SARS-COV-2 by Polymerase Chain Reaction (PCR) or as determined by clinical team

EXCLUSION CRITERIA:

1. Adults or Proxy unable to consent
2. Individuals who are not yet adults (infants, children, teenagers)
3. Pregnant women
4. Prisoners
5. Patients expected to die within 24 hours or with a "do not resuscitate" order,
6. Multi-organ failure,
7. History of hypersensitivity or allergy to any component of the study drug,
8. Ongoing massive surgical or unexplained bleeding,
9. History of bleeding or clotting disorder,
10. Severe traumatic brain injury (Glasgow Coma Scale <6),
11. Spinal or multiple-trauma,
12. Cancer (incurable/terminal phase) and/or patients receiving palliative care,
13. Enrollment in another concurrent clinical interventional study if considered interfering with this study objectives
14. Per study team discretion, any condition(s) that may prevent safe treatment, preclude adequate evaluation or adding further risk to their underlying illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Ginzburg, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker BM, Proctor KG, Guerra R, Manning RJ, Aguilar V, Meizoso JP, Pastewski A, Sneij W, Marttos AC, O'Neil CF, Ramsey WA, Namias N, Ginzburg E. A novel description of AT deficiency in hospitalized COVID-19 patients. Eur Rev Med Pharmacol Sci. 2025 Jan;29(1):30-38. doi: 10.26355/eurrev_202501_37057. PMID 39911044

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant death while on the study is considered completion of study.
Period: Screening Period
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Started | 20 | 20 | 12
Completed | 15 | 20 | 12
Not Completed | 5 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Participant discharged before receiving intervention | 3 | 0 | 0
Period: Treatment Period
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Started | 15 | 20 | 12
Completed | 15 | 20 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only | Total
Number analyzed (Participants) | 20 | 20 | 12 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 9 | 38
  >=65 years | 5 | 6 | 3 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 4 | 17
  Male | 14 | 13 | 8 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 14 | 7 | 31
  Not Hispanic or Latino | 10 | 6 | 5 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 4 | 17
  White | 12 | 14 | 8 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in ISTH DIC Score
Description: As measured by the International Society of Thrombosis and Haemostasis Disseminated Intravascular Coagulation scale (ISTH DIC) which has a total score ranging from 0-8 with a score of 5 and higher indicating overt DIC.
Time Frame: Baseline, Day 9
Population: Not all participants were able to complete the assessments required for evaluation of the DIC score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 15 | 12
score on a scale | 0.27 (1.71) | 0 (1.73) | 0 (1.65)

2. Secondary Outcome: Change in D-Dimer Levels
Description: D-Dimer levels assessed from blood samples will be evaluated in mcg/ml D-Dimer Units (DDU)
Time Frame: Baseline, Day 9
Population: Not all participants were able to complete the assessments required for the evaluation of the D-dimer.
Measure: Mean (Standard Deviation); unit: mcg/ml DDU
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 15 | 12
mcg/ml DDU | -1.97 (5.60) | 0.4 (3.18) | 0.25 (2.18)

3. Secondary Outcome: Change in Fibrinogen Levels
Description: Fibrinogen levels assessed from blood samples will be evaluated in mg/dL.
Time Frame: Baseline, Day 9
Population: Not all participants were able to complete the assessments required for evaluation of Fibrinogen levels.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 15 | 12
mg/dL | -102.1 (233.7) | -123 (215.1) | -111 (307.5)

4. Secondary Outcome: Change in Prothrombin Time
Description: Prothrombin time assessed from blood samples will be evaluated in seconds.
Time Frame: Baseline, Day 9
Population: Not all participants were able to complete the assessments required for evaluation of the Prothrombin Time levels.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 15 | 12
Seconds | 0.01 (2.07) | 0.31 (1.27) | 0.59 (1.39)

5. Secondary Outcome: Length of Hospital Stay
Description: Length of Hospital Stay reported in days.
Time Frame: Up to 60 days
Measure: Median (Standard Deviation); unit: Days
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 20 | 12
Days | 13 (15.1) | 6 (8.35) | 8.5 (9.46)

6. Secondary Outcome: Mortality Rate
Description: The number of participants with reported death.
Time Frame: Up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 20 | 12
Participants | 2 | 3 | 3

7. Secondary Outcome: Pulmonary Function
Description: Pulmonary Function will be reported as the mean days the participant was on any of the following: mechanical ventilation and/or Extracorporeal Membrane Oxygenation (ECMO) use.
Time Frame: Up to 60 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 20 | 12
Days | 1.33 (5.16) | 2.2 (6.70) | 3.08 (6.97)

8. Secondary Outcome: Change in SOFA Scores
Description: Sequential Organ Failure Assessment (SOFA) is scored from 0-4 with the higher score indicating more organ failure.
Time Frame: Baseline, Day9
Population: Not all participants were able to complete the assessments required for evaluation of the SOFA score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 14 | 15 | 12
score on a scale | 0.43 (3.41) | 1.23 (3.33) | 0.64 (2.27)

9. Secondary Outcome: Change in SOFA Respiratory Sub Score
Description: SOFA Respiratory Sub Score is scored from 0-4 with the higher score indicating worse organ failure.
Time Frame: Baseline, Day 9
Population: Not all participants were able to complete the assessments required for evaluation of the SOFA sub score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 15 | 12
score on a scale | -0.67 (0.98) | -0.07 (0.70) | -0.17 (1.69)

10. Secondary Outcome: Number of Events of Venous Thromboembolism
Description: Number of events of venous thromboembolisms from admission to hospital discharge.
Time Frame: Up to 60 days
Measure: Number; unit: Events
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 20 | 12
Events | 0 | 0 | 3

11. Secondary Outcome: Number of Events of Major Bleeding
Description: Number of events of major bleeding from admission to hospital discharge.
Time Frame: Up to 60 days
Measure: Number; unit: events
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 More Than 100% With SOC Only
Number analyzed (Participants) | 15 | 20 | 12
events | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: 60 days
Groups:
- AT3 Less Than 100% With SOC Plus AT3 Supplement: Participants in this group, with endogenous Antithrombin lll less than 100%, will receive up to 5 doses of supplemental Antithrombin III on Days 1, 3, 5, 7 and 9, in addition to standard of care (SOC) treatment.
  Antithrombin III: A daily dose from 1,821 to 9,100 IUs Antithrombin III, depending on participant's weight and current antithrombin II level, will be administered intravenously every other infusion day (Days 1, 3, 5, 7 and 9).
- AT3 of 100% or More, With SOC Only: Participants in this group, with endogenous Antithrombin III 100% or more, will receive SOC treatment only.
Arm/Group | AT3 Less Than 100% With SOC Plus AT3 Supplement | AT3 Less Than 100% With SOC Only | AT3 of 100% or More, With SOC Only
All-Cause Mortality (participants affected / at risk) | 2/15 | 3/20 | 3/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/20 | 0/12
Other Adverse Events (participants affected / at risk) | 5/15 | 5/20 | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AT3 Less Than 100% With SOC Plus AT3 Supplement (N=15) | AT3 Less Than 100% With SOC Only (N=20) | AT3 of 100% or More, With SOC Only (N=12)
Insomnia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 4 (4)
Shock (General disorders) | 1 (1) | 2 (2) | 2 (2)
Heart Failure with reduced Ejection Fraction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterovesical Junction (UVJ) Calculus (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Worsening Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 4 (4)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
Incidental Pulmonary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Necrotic Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Critical Illness Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asystole (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Bilateral Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated D-Dimer (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Severe Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Right Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous Emphysema w/ Pneumomdiastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dialysis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Thromocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Congestion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MSSA Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
With decreased Coronavirus disease of 2019 (COVID-19) cases, enrollment slowed leading to the early termination of the trial; the target number of 75 enrolled patients was not reached. Hesitancy to participate in the trial was noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT04899232/Prot_SAP_000.pdf